CLINICAL TRIAL: NCT05756426
Title: Consortium for Optimized Integration of Bio-Artificial Blood Components for Adaptive Resuscitation Therapy
Acronym: CONCERT
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Rogers, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP- 00104380
Record Dates: First submitted 2023-02-02; First posted 2023-03-06 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hemorrhage; Hemodynamic Instability
Keywords: Hemostasis; Vasoactivity; Oxygen affinity; Red Blood Cell; Whole blood analogue; Perfusion; Nitric Oxide; Methemoglobin
MeSH Terms: conditions — Hemorrhage | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Healthy Adult Volunteers: Healthy volunteers can be any adult, who meets eligibility criteria and is willing to donate blood for the purpose of this research study. The individual will have 20 milliliters (mL) of blood drawn upon the time of consent. The subject may donate up to 12 times (maximum) per year over the course of their enrollment, no closer together than every 2 weeks (14 days). Only basic demographic data will be collected (i.e., Age, Gender, Ethnicity, History of medical illness (or Primary Diagnosis), weight, and current medications/therapies). The Informed Consent Form Documentation Checklist & Specimen Collection Checklist will be utilized to ensure eligibility is checked and most recent Informed Consent Form (ICF) is signed prior to specimen collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers >/= 18yrs of age without acute or chronic illness.
  Interventions: Other: Prospective

INTERVENTIONS:
Other: Prospective — Single arm, healthy adult volunteers for blood donation.

SUMMARY:
There is need for a whole blood analog for use when banked blood is unavailable or undesirable.

In civilian trauma, hemorrhage accounts for ~ 35% of pre-hospital deaths; moreover, ~ 20% of military casualties are in hemorrhagic shock on arrival to field hospitals and an additional 5% require urgent transfusion. A recent review concluded that hemorrhage accounted for ~ 90% of potentially survivable battlefield deaths - lives that could be saved with better hemorrhage control capabilities and improved, field-ready blood, blood components, or blood substitutes. While study of ideal composition for resuscitative fluids is ongoing, it is evident that for those in hemorrhagic shock, volume replenishment alone (without O2 carrying capacity) is insufficient. Alternatively, with massive blood loss or with ongoing bleeding from non-compressible injuries, resuscitation with an O2 carrier alone may be complicated by acquired coagulopathy (either dilutional or trauma-induced).

Development of a balanced resuscitation fluid that treats both shock and coagulopathy (comprising a field-deployable O2 carrier with lyophilized humoral hemostatic components and platelets) is essential to allow on-scene treatment during the critical 'golden-hours' after injury. As such, the whole blood analog described herein could be this product, thus transforming care in both civilian and military settings.The scientific purpose of this study is to develop a combined whole blood substitute from individual artificial prototypes that have been separately developed for each blood component (i.e., combining an artificial oxygen carrier, with an artificial plasma analogue and an artificial platelet analogue). Together, these combined components will recapitulate the composition and performance of natural whole blood.

Blending and combination experiments of the individual artificial prototypes will be performed to test compatibility and optimize efficacy. State of the art in vitro (bench top) assays will be performed to assess physicochemical and functional performance (hemodynamics, oxygen delivery, hemostasis), with data being compared to experiments performed on fresh and stored whole blood.

DETAILED DESCRIPTION:
Previous blood substitutes have failed for 3 main reasons. (1) dysfunctional oxygen interactions resulting from fixed oxygen affinity, allowing adequate oxygen capture in the lungs, but poor oxygen release to tissue (i.e., oxygen affinity is not context responsive to physiologic cues of perfusion sufficiency such as pH, etc.), (2) interference with normal regulation of blood vessel caliber, with inappropriate trapping of the endogenous vasodilator nitric oxide resulting in intense vasoconstriction and tissue ischemia, and (3) inability to maintain hemoglobin functionality during circulation, with hemoglobin auto-oxidizing to methemoglobin which cannot carry and deliver oxygen, thus resulting in a drastically limited effective circulation time.

The individual artificial blood components, which will form the whole blood analog in this proposal, have been designed to overcome these previous design flaws. In addition, all components are amenable to facile reconstitution after extended, ambient dry storage, allowing sustained shelf stability.

In short, these components are ripe for integration to form a product recapitulating natural blood performance.

This study will use data and specimens collected under this protocol and will prospectively enroll new subjects at UMB for observational study. There will not be issues related to the probability of group assignment, the potential for subject to be randomized to a placebo group or the use of controlled substances.

There is only one cohort involved in this study

1. Prospective healthy adults (UMB only)

ELIGIBILITY:
Inclusion Criteria:

* Subject >/= 18 years of age
* Subject weighs >40kg (88lbs)
* Subject must be generally healthy

Exclusion Criteria:

* Suspected or diagnosed with ongoing (chronic) or acute infection
* Subject is pregnant
* Subject is non-english speaking

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research study intends to enroll 50healthy volunteer subjects/year over the next 5 years (total of 250 subjects).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Determine the hemoglobin based oxygen carrier (HBOC) amount in the whole blood analogue (WBA) that has the same oxygen delivery capacity as stored blood. | 4years
  Oxygen delivery capacity will be analyzed by measuring the oxygen disassociation curve and determining and arterial-venous (A-V) delta hemoglobin oxygen saturation. From this an A-V oxygen flux capacity can be determine and matched between stored blood and HBOC.
Evaluate performance attributes (PA's) stored whole blood (SWB): fresh whole blood, and WBA:fresh whole blood (FWB) mixtures. | 4years
  Compose mixtures of SWB:FWB or WBA:FWB, in ratios consistent of massive transfusions. Quantify (1) oxygen disassociation curve of mixtures across pH ranges of stressed physiology (pH 7.2-7.6). Determine the A-V delta hemoglobin saturation to calculate oxygen flux capacity. (2) viscosity shear relationships and visco elastic behavior will be characterized by rheometry, (3) Nitric oxide (NO) trapping and vasoactivity utilizing a biochemical NO trapping assay and a aortic rings (vascular ring bioassay), (4) hemostasis measuring thromboelastography (TEG).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rogers, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore (UMB), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided